CLINICAL TRIAL: NCT00754221
Title: A Multi-center, Long-term, Open-label Extension Study of [S,S]-Reboxetine (PNU-165442G) Administered Once Daily in Patients With Fibromyalgia
Brief Title: Open Label Extension Study of [S,S]-Reboxetine in Patients With Fibromyalgia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been terminated early as the esreboxetine development program is being discontinued. There are no safety or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6061053
Record Dates: First submitted 2008-09-16; First posted 2008-09-17 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Fibromyalgia
Keywords: Phase 3, safety study, [S,S]-Reboxetine, Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — O-methyl reboxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: [S,S]-Reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine — Once a day, oral treatment, of 4, 6, 8 or 10 mg

SUMMARY:
This is a study to investigate the long-term safety and effectiveness [S,S]-Reboxetine in relieving the symptoms of Fibromyalgia in patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, at least 18 years of age
* Patients must meet the ACR criteria for fibromyalgia (ie, widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites)
* Completed preceding double-blind randomized, controlled trial

Exclusion Criteria:

* Patients with other severe pain (eg, Diabetic Peripheral Neuropathy and PostHerpetic Neuralgia) that may confound assessment or self evaluation of the pain associated with fibromyalgia
* Patients with any autoimmune rheumatic disorder, non-focal rheumatic disease (other than fibromyalgia), active infection, or untreated endocrine disorder
* A current or recent diagnosis (last 6 months) or episode of major depressive disorder, dysthymia and/or uncontrolled depression
* History of mania, hypomania, other psychotic disorder, or current mood disorder with psychotic features

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Vital Signs | 66 weeks
12-Lead ECG | 66 weeks
Hematology & Biochemistry Laboratory Parameters | 66 weeks
Adverse Events | 66 weeks

SECONDARY OUTCOMES:
Short-Form 36 Health Survey | 66 weeks
Sheehan Disability Scale | 66 weeks
Pain Visual Analogue Scale | 66 weeks
Multidimensional Assessment of Fatigue | 66 weeks
Fibromyalgia Impact Questionaire | 66 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (98):
- United States (90):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Elk Grove, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Lafayette, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Winter Haven, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Gurnee, Illinois
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Mount Sterling, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Wheaton, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Wellesley Hills, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Edina, Minnesota
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Bend, Oregon
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Bridgeville, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Nassau Bay, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Ogden, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, Oregon, Wisconsin
- Canada (8):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Bathurst, New Brunswick
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061053&StudyName=Open%20label%20extension%20study%20of%20%5BS%2CS%5D-Reboxetine%20in%20patients%20with%20fibromyalgia